CLINICAL TRIAL: NCT02729272
Title: Ultrasonic Versus Monopolar Energy-based Surgical Device in Colpotomy During Total Laparoscopic Hysterectomy in Terms of Surgical Smoke and Lateral Thermal Damage: a Randomized Controlled Trial (ULMOST Trial)
Brief Title: Ultrasonic Versus Monopolar Energy-based Surgical Device in Colpotomy
Acronym: ULMOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-04-012
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Gynecologic Diseases
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonic ESD (Experimental): Laparoscopic colpotomy by ultrasonic ESD (Harmonic Synergy Hook Blade; Ethicon Endo-Surgery) during total laparoscopic hysterectomy.
  Interventions: Procedure: Laparoscopic colpotomy by ultrasonic ESD; Device: Ultrasonic ESD
- Monopolar ESD (Active Comparator): Laparoscopic colpotomy by monopolar ESD (hook electrode with 90 watts of unmodulated current; Karl Storz, Tuttlingen, Germany) during total laparoscopic hysterectomy.
  Interventions: Procedure: Laparoscopic colpotomy by monopolar ESD; Device: Monopolar ESD

INTERVENTIONS:
Procedure: Laparoscopic colpotomy by ultrasonic ESD — In this intervention, laparoscopic colpotomy was performed by ultrasonic ESD (Harmonic Synergy Hook Blades; Ethicon Endo-Surgery, Cincinnati, OH, USA).
  Arms: Ultrasonic ESD
Procedure: Laparoscopic colpotomy by monopolar ESD — In this intervention, laparoscopic colpotomy was performed by monopolar ESD (hook electrode with 90 watts of unmodulated current; Karl Storz, Tuttlingen, Germany).
  Arms: Monopolar ESD
Device: Monopolar ESD
  Arms: Monopolar ESD
Device: Ultrasonic ESD
  Arms: Ultrasonic ESD

SUMMARY:
The aim of this randomized trial was to compare the degree of surgical smoke obstructing vision and thermal damage caused by two different ESDs (ultrasonic versus monopolar ESD) in colpotomy during total laparoscopic hysterectomy.

DETAILED DESCRIPTION:
According to previous studies performed in porcine and bovine tissues, ultrasonic energy based surgical devices (ESDs) created less surgical smoke, involved less visual obstruction, and produced less lateral thermal damage than monopolar ESDs. However, there was no study comparing ultrasonic ESD and monopolar ESD in laparoscopic colpotomy in terms of surgical smoke and lateral thermal damage. Therefore, the aim of this randomized trial was to compare the degree of surgical smoke obstructing vision and thermal damage caused by two different ESDs (ultrasonic versus monopolar ESD) in colpotomy during total laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* women with gynecologic diseases, such as uterine myoma, adenomyosis, and ovarian tumor;
* women who were planning to undergo TLH;
* women between 19 and 75 years of age.

Exclusion Criteria:

* women with any suggestion of malignant cervical or vaginal pathologies
* women with uncontrolled medical comorbidities or psychiatric illness, which could affect follow-up and/or compliance
* women who refused to participate or give consent to the procedures.

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Degree of surgical smoke obstructing vision | Day of surgery
  The degree of surgical smoke obstructing laparoscopic view was assessed by an independent, blinded, gynecologic surgeon who reviewed videotapes of each patient's laparoscopic colpotomy procedure using a 5-point Likert scale (1 = very clear; 2 = quite clear; 3 =somewhat smoky; 4 = quite smoky; and 5 = extremely smoky), and a higher score indicates a worse visuality
Degree of lateral thermal damage | Day of surgery
  Using a light microscope, the width of lateral thermal damage was measured from the point of instrument application to the margins of unchanged nearby tissue

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD,PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, NJ, South Korea

IPD SHARING:
Plan to Share IPD: No